CLINICAL TRIAL: NCT00540826
Title: Treatment Adherence and Compliance in Children and Adolescents on ADHD Medication and Emotional Expression in Clinical Practice
Brief Title: Treatment Compliance in Children and Adolescents on ADHD Medication
Acronym: COMPLY
Status: Completed | Type: Observational
Sponsor: Eli Lilly and Company (Industry)
Other Study IDs: 12067; B4Z-SB-B012
Record Dates: First submitted 2007-10-05; First posted 2007-10-08 (Estimated); Last update posted 2009-08-27 (Estimated); Status verified 2009-08

CONDITIONS: ADHD
MeSH Terms: conditions — Attention Deficit Disorder with Hyperactivity | interventions — Atomoxetine Hydrochloride; Central Nervous System Stimulants

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No

GROUPS / COHORTS (2):
- A: A: ADHD-patients receiving non-stimulants (e.g. atomoxetine)
  Interventions: Drug: Atomoxetine
- B: B: ADHD-patients receiving stimulants
  Interventions: Drug: stimulants (any approved ADHD medication)

INTERVENTIONS:
Drug: Atomoxetine — in-label use
  Other Names: Strattera
  Groups: A
Drug: stimulants (any approved ADHD medication) — in-label use
  Groups: B

SUMMARY:
The primary research objective of this observational study is to evaluate treatment compliance over one year in children and adolescents who are newly initiated on medication approved for the treatment of ADHD in a routine clinical setting. Compliance will be assessed using the Pediatric Compliance Self-Rating (PCSR) Instrument. A patient will be considered as compliant at a given visit, if the PCSR score is at least 5, corresponding to taking the medication at least often.

ELIGIBILITY:
Inclusion Criteria:

* 6-17 years old
* diagnosis of ADHD according to ICD-10 or DSM-IV criteria
* new initiation onto an approved medication to treat ADHD

Exclusion Criteria:

* no specific exclusion criteria

Ages: 6 Years to 17 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child
Study Population: Children and adolescents who are newly initiated on medication approved for the treatment of ADHD in a routine clinical setting.
  Participating physicians may be office or hospital based psychiatrists and pediatricians throughout Germany.
Sampling Method: Non-Probability Sample
Enrollment: 518 (Actual)
Dates: Start 2007-11; Study Completion 2009-06 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Call 1-877-CTLILLY (1-877-615-4559) or 1-317-615-4559 Mon-Fri 9 AM to 5 PM Eastern Time (UTC/GMT - 5 hours, EST), Study Director — Eli Lilly and Company
Locations (1):
- For additional information regarding investigative sites for this trial, contact 1-877-CTLILLY (1-877-285-4559, 1-317-615-4559) Mon - Fri from 9 AM to 5 PM Eastern Time (UTC/GMT - 5 hours, EST), or speak with your personal physician., Bad Homburg, Germany

REFERENCES:
- [Derived] Dittmann RW, Banaschewski T, Schacht A, Wehmeier PM. Findings from the observational COMPLY study in children and adolescents with ADHD: core symptoms, ADHD-related difficulties, and patients' emotional expression during psychostimulant or nonstimulant ADHD treatment. Atten Defic Hyperact Disord. 2014 Dec;6(4):291-302. doi: 10.1007/s12402-014-0136-z. Epub 2014 Apr 6. PMID 24705867
- See also: Lilly Clinical Trial Registry — http://lillytrials.com